CLINICAL TRIAL: NCT05096299
Title: OCS Heart EXPAND + CAP Continued Follow-Up Post-Approval Study
Brief Title: OCS Heart EXPAND + CAP Continued Follow-Up
Status: Active, not recruiting | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCS-HEART-02-PAS
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Heart Transplant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: OCS Heart — Transplanted with OCS preserved heart.

SUMMARY:
Post-approval observational study of subjects that were enrolled and transplanted in the OCS Heart EXPAND and OCS Heart EXPAND CAP studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients transplanted in the OCS Heart EXPAND and EXPAND CAP trials

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients transplanted in the OCS Heart EXPAND and EXPAND CAP trials will comprise the patient population for this PAS.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Patient survival | 5 years post transplant
  Patient survival through 5 years post-transplant

OTHER OUTCOMES:
Cardiac patient survival | 5 years post transplant
  Cardiac related patient survival through 5 years post-transplant
Graft survival | 5 years post transplant
  Graft survival through 5 years post-transplant